CLINICAL TRIAL: NCT04227626
Title: A Feasibility Study of Automated Glucose Control With the Gen2 GlucoSTAT Bionic Pancreas in Volunteers With Type 1 and Type 2 Diabetes
Brief Title: Inpatient Closed Loop Glucose Control With the Gen 2 GlucoSTAT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has not started, the device is not ready so the study will be delayed
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beta Bionics, Inc. (Industry)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P000079
Record Dates: First submitted 2020-01-10; First posted 2020-01-13 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes Treated With Insulin
Keywords: closed loop; insulin; dextrose
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- GlucoSTAT (Experimental): Type 1 diabetes and Type 2 diabetes with a total daily dose (TDD) of insulin that is > 0.75 u/kg or ≥ 2 u/kg.
  Interventions: Device: GlucoSTAT

INTERVENTIONS:
Device: GlucoSTAT — Closed-loop blood glucose control using intravenous insulin and dextrose
  Other Names: Closed-loop blood glucose control

SUMMARY:
The goal of this study is to perform a first-in-humans trial of a fully integrated, automated, closed-loop blood glucose control system designed for inpatient use. The GlucoSTAT was designed for use by patients with diabetes while they are in the hospital, and others who may develop high blood sugar as a result of their medical problems.

DETAILED DESCRIPTION:
Our envisioned end product is an in-patient automated closed-loop control system for PG regulation in the ICU as well as on the general hospital wards. In order to qualify the system for the broad spectrum of challenges it will face in the inpatient setting, this study will test the ability of the new integrated configuration of the system (the GlucoSTAT) to control PG in subjects with extremes of insulin sensitivity. The first goal of this study is to test the safety and efficacy of the control system in insulin sensitive subjects with type 1 diabetes. The second goal of this study is to test the safety and efficacy of the control system in subjects with type 2 diabetes and substantial insulin resistance (TDD > 0.75 u/kg/day, with up to 3 subjects with a TDD > 2 u/kg/day).

ELIGIBILITY:
Inclusion Criteria:

Type 1 diabetes:

1. Age 18 years or older with clinical type 1 diabetes for at least one year.
2. Diabetes currently managed using an insulin infusion pump and rapid- or very-rapid-acting insulins including insulin aspart (NovoLog or Fiasp), insulin lispro (Humalog), and insulin glulisine (Apidra).
3. Total daily dose (TDD) of insulin that is ≤ 1 U/kg
4. Prescription medication regimen stable for at least 1 month.
5. Informed consent obtained before any trial-related activities.

Type 2 diabetes:

1. Age 18 years or older with clinical type 2 diabetes for at least 1 year.
2. Diabetes currently managed using NPH as the basal insulin, which may be supplemented with regular or rapid-acting insulin and/or other anti-diabetic drugs.
3. Total daily dose (TDD) of insulin that is > 0.75 u/kg

   * Our goal is to have up to 3 T2D subjects with a TDD > 2 u/kg
4. Prescription medication regimen stable for at least 1 month.
5. Informed consent obtained before any trial-related activities.

Exclusion Criteria:

1. Unable to provide informed consent.
2. Unable to comply with study procedures.
3. Current participation in another diabetes-related clinical trial that, in the judgement of the principal investigator, will compromise the results of this study or the safety of the participant
4. Use of a long-acting insulin (in type 1 diabetes subjects) or a long-acting insulin other than NPH (in type 2 diabetes subjects), including insulin glargine (Lantus), insulin detemir (Levemir), insulin degludec (Tresiba), or ultra-lente.
5. Pregnancy (positive urine HCG), breast feeding, plan to become pregnant in the immediate future, or sexually active without use of contraception.
6. Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to RF interference.
7. Established history of latex, adhesive, or tape allergy that must be used in the study
8. Inadequate venous access as determined by study nurse or physician at time of screening.
9. Employed by, or having immediate family members employed by Beta Bionics, or being directly involved in conducting the clinical trial, or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial.
10. A condition that in the opinion of the investigator could interfere with the safe completion of the study. Conditions to be considered by the investigator may include the following:

    * Alcohol or drug abuse
    * Use of prescription drugs that may dull the sensorium, reduce sensitivity to symptoms of hypoglycemia, or hinder decision making during the period of participation in the study
    * Renal failure
    * Coronary artery disease that is not stable with medical management, including unstable angina, angina that prevents moderate exercise (e.g. climbing a flight of stairs) despite medical management, or within the last 12 months before screening a history of myocardial infarction, percutaneous coronary intervention, enzymatic lysis of a presumed coronary occlusion, or coronary artery bypass grafting
    * Congestive heart failure with New York Heart Association (NYHA) Functional Classification III or IV
    * History of TIA or stroke in the last 12 months
    * Untreated or inadequately treated mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Average plasma glucose over the closed-loop control period | every 15 minutes for 8.5 hours
  Average plasma glucose

SECONDARY OUTCOMES:
Number of carbohydrate interventions needed to treat hypoglycemia | 8.5 hour experiment duration
  The number of times that carbohydrates were consumed in response to hypoglycemia throughout the 8.5 hour experiment
Grams of carbohydrates needed to treat hypoglycemia | 8.5 hour experiment duration
  The amount of carbohydrates consumed in response to hypoglycemia throughout the 8.5 hour experiment
Carbohydrate content and total calories of consumed lunch meal | during 30 minute meal
  The amount of carbohydrates and total calories the subject consumed during their provided lunch
Insulin dosing (u/kg) | 8.5 hour experiment duration
  Total amount of insulin delivered by the GlucoSTAT during the experiment
Dextrose dosing (g/kg) | 8.5 hour experiment duration
  Total amount of dextrose delivered by the GlucoSTAT during the experiment

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States